CLINICAL TRIAL: NCT02258152
Title: SYN120 a Dual 5-HT6/5-HT2A Antagonist Proof of Concept Study to Evaluate Its Safety, Tolerability and Efficacy in Parkinson's Disease Dementia (SYNAPSE)
Brief Title: SYN120 Study to Evaluate Its Safety, Tolerability and Efficacy in Parkinson's Disease Dementia (SYNAPSE)
Acronym: SYNAPSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Massachusetts General Hospital (Other); Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYN120-CL03
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease Dementia (PDD)
Keywords: PDD; Parkinson's Disease Dementia; patients taking a cholinesterase inhibitor.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SYN120 (Experimental)
  Interventions: Drug: SYN120

INTERVENTIONS:
Drug: SYN120 — SYN120 Doses to be Administered: 20 mg QD (1 week titration), 50 mg QD (1 week titration), 100 mg QD (14 weeks of maintenance).
  Arms: SYN120
Drug: Placebo — Placebo QD
  Arms: Placebo

SUMMARY:
The purpose of this study placebo-controlled, randomized, double-blind study is to assess the safety and efficacy of SYN120 in patients with Parkinson's disease dementia (PDD) already treated with a stable dose of a cholinesterase inhibitor.

DETAILED DESCRIPTION:
This study includes a Screening Period of up to 6 weeks, a 16 week Treatment Period, and a 2 week Safety Follow Up Period.

Final eligibility will be determined at the Baseline Visit. Eligible patients will be randomized to receive placebo or SYN120 100 mg once a day (QD).

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease Dementia
* Patient has a routine caregiver
* Taking a stable cholinesterase inhibitor.
* Patient has a Montreal Cognitive Assessment (MoCA) 10-23 inclusive

Exclusion Criteria:

* History of any significant neurologic or psychiatric disease other than PD
* Any other condition or clinically significant abnormal findings that would make the patient unsuitable for the study
* Unpredictable motor fluctuations that would interfere with administering assessments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kenney, Study Director — Acorda Therapeutics
Locations (20):
- United States (20):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Sun Health Research Institute, Sun City, Arizona
  - UC San Diego, La Jolla, California
  - Parkinson's Disease & Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Carver College of Medicine, Iowa City, Iowa
  - Parkinson's Disease & Movement Disorder Center, University of Kansas Medical Center, Kansas City, Kansas
  - Department of Neurology, University of Maryland Parkinson's Disease & Movement Disorder Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Atlantic Neuroscience Institute, Summit, New Jersey
  - Duke University, Durham, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - Parkinson's Disease Movement Disorder Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Univeristy, Houston, Texas
  - Houston Methodist Neurological Institute/Movement Disorders Clinic, Houston, Texas

REFERENCES:
- [Derived] Fernandez HH, Weintraub D, Macklin E, Litvan I, Schwarzschild MA, Eberling J, Videnovic A, Kenney CJ; Parkinson Study Group SYNAPSE Investigators. Safety, tolerability, and preliminary efficacy of SYN120, a dual 5-HT6/5-HT2A antagonist, for the treatment of Parkinson disease dementia: A randomized, controlled, proof-of-concept trial. Parkinsonism Relat Disord. 2023 Sep;114:105511. doi: 10.1016/j.parkreldis.2023.105511. Epub 2023 Jul 13. PMID 37532622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 18 study centers in the US. Combined, a total of 82 patients were randomized: 44 patients to treatment with placebo and 38 to treatment with SYN120, 100 mg QD (once a day). Of these patients, 72 (88%) completed the study.
Period: Overall Study
Arm/Group | Placebo | SYN120
Started | 44 | 38
Completed | 38 | 34
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Population: The Safety Population (safety analysis set) consisted of patients who received a dose of placebo or SYN120; all 82 patients randomized in this study were included in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SYN120 | Total
Number analyzed (Participants) | 44 | 38 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 41 | 31 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.13 (5.86) | 72.13 (8.13) | 73.21 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 41 | 32 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 37 | 81
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 43 | 38 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 38 | 82
Weight at Screening [Mean (Standard Deviation); unit: kg] | 81.03 (16.31) | 76.54 (10.69) | 78.95 (14.09)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Objective of This Study is to Assess the Efficacy of SYN120 on Cognition as Determined by the Cognitive Drug Research Computerized Cognition Battery (CDR) Continuity of Attention in Patients With Parkinson's Disease.
Description: To access the effect of SYN-120 for Continuity of Attention, a measure which reflects the ability to sustain attention and avoid error The Cognitive Drug Research Computerized Cognition Battery is a computerized neuropsychological test battery to assess cognitive tasks based on measures of Vigilance (1 - 180 seconds) and Choice Reaction Time (1 - 120 seconds). The stimuli are presented on a computer screen and the subjects respond by pressing either a "Yes" or "No" on a response box. It is a time measured test.
  The ability to keep mind on a single task over time. COA is calculated as (VIGACC*0.45) + (CRTACC*0.5) - where VIGACC is digit vigilance accuracy, CRTACC is choice reaction time accuracy. Higher COA scores represent greater sustained attention and avoidance of errors.
Time Frame: up to Week 16
Population: Protocol Deviation: No patient was discontinued from the study due to a protocol deviation and results based on the PP (per-protocol analysis set) population are similar to those from the mITT (modified intention-to-treat analysis set) population. Patients were not withdrawn from the study despite meeting withdrawal criteria.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | SYN120
Number analyzed (Participants) | 38 | 34
Seconds
  Screening (1) | 77.04 (15.56) | 75.61 (21.39)
  Screening (2) | 80.97 (13.66) | 80.70 (16.80)
  Baseline | 80.95 (11.45) | 80.98 (13.01)
  Week 8 | 78.83 (17.08) | 77.68 (19.60)
  Week 16 | 81.25 (12.36) | 79.37 (15.90)
  Change from Week 0 to 8 | -1.88 (16.73) | -3.31 (12.22)
  Change from Week 0 to 16 | -0.35 (10.51) | -3.70 (12.86)

2. Secondary Outcome: To Assess the Effects of SYN120 on Cognitive Drug Research Computerized Cognition Battery (CDR) Quality of Episodic Memory (QEM)
Description: To access the effects of SYN120 for Quality of Episodic Memory. QEM measures the ability to store, hold, and retrieve information of an episodic nature. The stimuli are presented on a computer screen and the subjects respond by pressing either a "Yes" or "No" on a response box. It is a time measured test.
  Quality of Episodic Memory is calculated as (DRECOACC + DRECNACC - 100) + (DPICOACC + DPICNACC - 100) +((IRCL - IRCLERR)*100 / 15) + ((DRCL - DRCLERR)*100 / 15), where DRECOACC is Word Recognition original stimuli accuracy (1 - 120 seconds), DRECNACC is word recognition new stimuli accuracy, DPICOACC is Picture Recognition original stimuli accuracy (1 - 120.5 seconds), DPICNACC is picture recognition new stimuli accuracy, IRCL is Immediate Word Recall (1 - 120.5 seconds), IRCLERR is immediate word recall errors, DRCL is Delayed Word Recall (1 - 120.5 seconds), and DRCLERR is delayed word recall errors. Higher QEM scores greater ability to retain memory.
Time Frame: up to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | SYN120
Number analyzed (Participants) | 38 | 34
Seconds
  Screening (1) | 107.66 (55.49) | 116.14 (60.50)
  Screening (2) | 111.98 (55.62) | 99.69 (30.11)
  Baseline | 117.70 (49.68) | 114.13 (45.93)
  Week 8 | 123.58 (52.03) | 118.37 (61.95)
  Week 16 | 112.43 (69.50) | 118.20 (54.08)
  Change from Week 0 to 8 | 5.89 (46.66) | 4.25 (49.02)
  Change from Week 0 to 16 | -5.77 (55.41) | -0.08 (45.33)

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: Safety evaluation was based on the Safety Population which included all 82 patients enrolled into the study.
Arm/Group | Placebo | SYN120
All-Cause Mortality (participants affected / at risk) | 0/44 | 1/38
Serious Adverse Events (participants affected / at risk) | 5/44 | 4/38
Other Adverse Events (participants affected / at risk) | 34/44 | 28/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | SYN120 (N=38)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | SYN120 (N=38)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 7 (8)
Fall (Injury, poisoning and procedural complications) | 8 (12) | 5 (5)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Haemoglobin Decreased (Investigations) | 2 (2) | 2 (2)
Cognitive Disorder (Nervous system disorders) | 3 (3) | 2 (4)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (4)
Confusional State (Psychiatric disorders) | 5 (5) | 4 (4)
Hallucination, Visual (Psychiatric disorders) | 2 (2) | 5 (5)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT02258152/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT02258152/SAP_001.pdf